CLINICAL TRIAL: NCT05811000
Title: A Phase 2 Clinical Study to Explore the Optimal Dosage/Administration of PM012 Tablet in Alzheimer's Disease: Double-Blind, Randomized Between Placebo Control Group and Dose Groups, Parallel-Design, Multicenter Study
Brief Title: A Phase 2 Clinical Study to Explore the Optimal Dosage/Administration of PM012 Tablet in Alzheimer's Disease
Acronym: PM012-2b
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mediforum Ltd., Co. (Industry)
Collaborators: LSK Global Pharma Services Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MFDS-31834
Record Dates: First submitted 2023-03-17; First posted 2023-04-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Mild Alzheimer Disease
Keywords: Alzheimer's Disease; Dementia; Brain Diseases; Central Nervous System Disease; Nervous System Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aricept 5 mg (Active Comparator): Aricept 5 mg + Placebo of PM012 eight tablets, daily during 12 weeks (oral)
  Interventions: Drug: PM012 Placebo; Drug: Donepezil
- PM012 2,600 mg (Experimental): PM012 2,600 mg + Placebo of PM012 four tablets +Placebo of Aricept one tablet, daily during 12 weeks (oral)
  Interventions: Drug: PM012; Drug: PM012 Placebo; Drug: Donepezil placebo
- PM012 3,900 mg (Experimental): PM012 3,900 mg + Placebo of PM012 two tablets +Placebo of Aricept one tablet, daily during 12 weeks (oral)
  Interventions: Drug: PM012; Drug: PM012 Placebo; Drug: Donepezil placebo
- PM012 5,200 mg (Experimental): PM012 5,200 mg + Placebo of Aricept one tablet, daily during 12 weeks (oral)
  Interventions: Drug: PM012; Drug: Donepezil placebo

INTERVENTIONS:
Drug: PM012 — PM012 650 mg tablet drug
  Arms: PM012 2,600 mg; PM012 3,900 mg; PM012 5,200 mg
Drug: PM012 Placebo — PM012 tablet placebo
  Arms: Aricept 5 mg; PM012 2,600 mg; PM012 3,900 mg
Drug: Donepezil — Aricept 5 mg (donepezil hydrochloride) drug
  Arms: Aricept 5 mg
Drug: Donepezil placebo — Aricept 5 mg (donepezil hydrochloride) placebo
  Arms: PM012 2,600 mg; PM012 3,900 mg; PM012 5,200 mg

SUMMARY:
To evaluate the safety and efficacy of PM012 tablets for Alzheimer's disease, dose-finding study will be performed on phase 2b, and the established dose will be used for the non-inferiority phase 3 trial to evaluate the investigational product's safety and efficacy: Double blind, randomized, active drug comparative, multi-center, parallel-group clinical trial

DETAILED DESCRIPTION:
This study is to establish an effective therapeutic dose in Korean patients with a mild degree of Alzheimer's disease, by comparing the safety and efficacy of the investigational product PM012 tablet administered to the 2,600 mg /day group, 3,900 mg /day group, and 5,200 mg /day group, with the active drug Aricept 5 mg (donepezil hydrochloride) from Daewoong Pharmaceuticals administered to the active control group, for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1) Male and female patients aged ≥ 50 and ≤ 85 years.
* 2) Patients clinically diagnosed as probable Alzheimer's disease based on DSM-IV and NINCDS-ADRDA criteria.
* 3) Patients between MMSE score of 20~26 at screening visit.
* 4) Patients with Global CDR score of 0.5 or 1 at the screening visit.
* 5) Patients administered with donepezil 5㎎ stably for over 3 months or who have never been administered donepezil.
* 6) Patients who can perform cognitive or other necessary tests.
* 7) Patients who have a caretaker who can accompany the patient for all clinical visits and for the primary efficacy evaluation (a caretaker is a family member or someone trustworthy who provides care for daily activities, spending more than 8 hours per week with patients).
* 8) Patients who have consented to participate in medically acceptable contraception*

  * Effective contraception methods: Infertility surgery of the patient or his/her spouse (vasectomy, tubal ligation), placement of an intrauterine contraceptive device, double barrier method (concomitant use of spermicides and condoms, and contraceptive diaphragms, vaginal sponges, or cervical caps). Oral contraceptives and intermittent celibacy (absolute celibacy is allowed) are not acknowledged as effective contraceptive methods.
* 9) Patients who have signed the informed consent on his/her own will

Exclusion Criteria:

* 1) Patients with hypersensitivity to the investigational product or components contained in the investigational product.
* 2) Patients with hypersensitivity to piperidine derivatives.
* 3) Patients with possible, probable or definite vascular dementia according to the NINDS-AIREN criteria.
* 4) History (cerebrovascular disease, structural or developmental malformations, epilepsy, contagious, degenerative, or infectious/demyelinating CNS status) and/or evidence (CT or MRI results performed at screening or within 12 months) of other CNS diseases as the major cause of dementia.
* 5) Patients who are illiterate.
* 6) Patients with severe hearing or visual disabilities so that efficacy assessment is impossible.
* 7) Abnormal test results for vitamin B12, serologic testing for syphilis, or thyroid stimulating hormone (TSH) that may have contributed to or may be the cause of patient's dementia.
* 8) Patients with a history of significant psychiatric disease such as schizophrenia or bipolar disorder that may interfere with participation in the trial as viewed by the investigator, or patients with current major depression disorder (Short Form GDS ≥ 7) (However, patients who depressed due to Alzheimer's disease can participate in this trial by the investigator).
* 9) Patients with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* 10) Patients with a history of known or suspected seizure including febrile seizure, or recent history of loss of consciousness or a history of significant head trauma with loss of consciousness.
* 11) Patients with gastrointestinal, endocrinological, or cardiovascular disorders that is not controlled by diet or drugs.
* 12) Patients with cardiac diseases such as myocardial infarction, valvular heart disease, or arrhythmia within 3 months prior to screening.
* 13) Patients with asthma or obstructive pulmonary diseases that is not controlled by drugs.
* 14) Patients with extrapyramidal disorders (Parkinson's disease, Parkinsonism, etc).
* 15) Patients with dementia due to Creutzfeldt-Jakob disease, Pick's disease, or Huntington's disease.
* 16) Patients with uncontrolled diabetes (HbA1c > 8.0%) or insulin dependent diabetes.
* 17) Patients with a history of alcohol or other substance abuse.
* 18) Patients with hypertension with systolic pressure over 165mmHg or diastolic pressure over 96mmHg.
* 19) Patients with severe renal dysfunction (Serum creatinine over 2.0㎎/dl).
* 20) Patients with severe liver dysfunction (ALT, AST, total bilirubin more than 2.5-fold the upper normal limit).
* 21) Patient who has been administered drugs that Dementia drugs(Donepezil, Galantamine, Memantine, Rivastigmine tartrate) within 3 months prior to screening (However, patients who have been administered donepezil 5mg stably for over 3 months are excluded).
* 22) Patient who has required to take restricted drugs other than investigational products during the clinical trial period.
* 23) patient who has unabled to take concomitant drugs during the clinical trial period under the following conditions : It was taken without dose change 2 months before randomization, and was taken without dose change during the clinical trial period (except for drugs allowed to be taken as needed).
* 24) Patients with a history of clinically significant drug hypersensitivity reaction.
* 25) Patients who have been administered investigational products from another clinical trial within 3 months prior to participation in this trial.
* 26) Patients who are deemed unfit to participate in this trial by the investigator.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2024-08-13 (Estimated)

PRIMARY OUTCOMES:
ADAS-cog (Alzheimer's Disease Assessment Scale-cognitive subscale) | At 12 weeks post-dose
  * To compare the efficacy of dose groups and active comparator group based on cognitive functions assessed through ADAS-cog at 12 weeks post-dose.
  * The total score ranges from 0 (no function) to 70 (maximal function), and the higher the score, the greater the cognitive impairment.
ADCS-MCI-ADLI (Alzheimer's Disease Cooperative Study-Mild Cognitive Impairment- Activities of Daily Living Inventory) | At 12 weeks post-dose
  * To compare the efficacy of dose groups and active comparator group based on activities of daily living assessed through ADCS-MCI-ADLI at 12 weeks post-dose
  * The total score ranges from 0 to 53, and the lower the score, the more the participant needs help with daily living.

SECONDARY OUTCOMES:
ADAS-cog (Alzheimer's Disease Assessment Scale-cognitive subscale) | At 8 weeks post-dose
  * To compare the efficacy of dose groups and active comparator group based on cognitive functions assessed through ADAS-cog at 8 weeks post-dose.
  * The total score ranges from 0 (no function) to 70 (maximal function), and the higher the score, the greater the cognitive impairment.
ADCS-MCI-ADLI (Alzheimer's Disease Cooperative Study-Mild Cognitive Impairment-Activities of Daily Living Inventory) | At 8 weeks post-dose
  * To compare the efficacy of dose groups and active comparator group based on activities of daily living assessed through ADCS-MCI-ADLI at 8 weeks post-dose.
  * The total score ranges from 0 to 53, and the lower the score, the more need to help with daily living.
CDR (Clinical Dementia Rating) | At 8 weeks and 12 weeks post-dose
  * To compare the efficacy of dose groups and active comparator group based on overall function assessed through CDR at 8 weeks and 12 weeks post-dose.
  * Scores are on a scale of 0 - 5, with 0 = no dementia, 0.5 = questionable dementia, 1 = mild dementia, 2 = moderate dementia, 3 = severe dementia, 4 = profound dementia, and 5 = terminal dementia.
MMSE (Mini Mental State Examination) | At 8 weeks and 12 weeks post-dose
  * To compare the efficacy of dose groups and active comparator group based on cognitive functions assessed through MMSE at 8 weeks and 12 weeks post-dose.
  * The total score ranges from 0 to 30 and the lower the score, the more the cognitive problems.
NPI (Neuropsychiatric Inventory) | At 8 weeks and 12 weeks post-dose
  * To compare the efficacy of dose groups and active comparator group based on behavioral change assessed through NPI at 8 weeks and 12 weeks post-dose.
  * The total score ranges from 0 to 144 and the higher the score, the more neuropsychiatric symptoms.
Number of participants with adverse events, with abnormal physical exam findings and abnormal laboratory tests results. | At 12 weeks post-dose
  - To compare the safety of dose groups and active comparator group based on adverse events and clinical laboratory tests at 12 weeks post-dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Mediforum, Seoul, Seongdon-gu, South Korea

REFERENCES:
- See also: Safety and efficacy assessment of standardized herbal formula PM012 — https://pubmed.ncbi.nlm.nih.gov/22458507/
- See also: Standardized Herbal Formula PM012 Decreases Cognitive Impairment and Promotes Neurogenesis in the 3xTg AD Mouse Model of Alzheimer's Disease — https://pubmed.ncbi.nlm.nih.gov/26446019/